CLINICAL TRIAL: NCT03908177
Title: Comparative Performance of Zirconia Tissue Level Implants vs. Titanium Bone Level Implants Placed With a Fully Digital Workflow: A Multicentre Multinational Randomized Controlled Clinical Trial
Brief Title: Comparison of Clinical Performance and Safety of Zirconia vs. Titanium Implants: a Multi-national RCT.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Straumann AG (Industry)
Collaborators: Avania (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR2017-04
Record Dates: First submitted 2019-04-05; First posted 2019-04-09 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-05

CONDITIONS: Dental Implants, Single-Tooth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Group (SG) (Experimental): Receive new zirconia implant: Straumann® PURE 2-piece Ceramic Implant (tissue level), ZLA
  Interventions: Device: Ceramic Dental Implant
- Control Group (CG) (Active Comparator): Receive standard titanium implant: Straumann® Bone Level Implant, Titanium, SLA
  Interventions: Device: Titanium Dental Implant

INTERVENTIONS:
Device: Ceramic Dental Implant — The ceramic implant will be placed in healed extraction sockets in the premolar-to-premolar area in the mandible and maxilla for single tooth replacement followed by prosthetic loading after 4 months healing time. Type 4 surgery will be performed as defined by the ITI Consensus Statements for Implant Placement in Extraction Sockets: healed sites, typically around 16 weeks after tooth was extracted or after tooth was lost to allow complete healing of the ridge as well as soft- and hard tissue maturation. Both SG and CG receive routine treatment, only the choice of the implant material is defined by the study protocol.
  Arms: Study Group (SG)
Device: Titanium Dental Implant — The titanium implant will be placed in healed extraction sockets in the premolar-to-premolar area in the mandible and maxilla for single tooth replacement followed by prosthetic loading after 4 months healing time. Type 4 surgery will be performed as defined by the ITI Consensus Statements for Implant Placement in Extraction Sockets: healed sites, typically around 16 weeks after tooth was extracted or after tooth was lost to allow complete healing of the ridge as well as soft- and hard tissue maturation. Both SG and CG receive routine treatment, only the choice of the implant material is defined by the study protocol.
  Arms: Control Group (CG)

SUMMARY:
A post-market, multi-centre, prospective, open, randomized-controlled, non-inferiority clinical study to compare short-term performance and safety of the Straumann PURE 2-piece Ceramic Implant with Straumann Bone Level Implant using a fully digital workflow.

DETAILED DESCRIPTION:
To compare short-term performance and safety of the Straumann PURE 2-piece Ceramic Implant with Straumann Bone Level Implant using a fully digital workflow. Post-market, multi-centre, prospective, open, randomized-controlled, non-inferiority clinical study investigating patients in need of dental implant therapy for single-tooth gap rehabilitation. The follow up time is1 year after final crown restoration.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have voluntarily signed the Informed Consent Form before any study related procedures are performed, are willing and able to attend scheduled follow-up visits and agree that the pseudonymized data will be collected, analysed, and published.
* Patients must be males or females who are a minimum of 18 years of age.
* Patients, who are in need of a single tooth replacement with a dental implant in the premolar-to-premolar area in the mandible or maxilla (excluding lower incisors).
* Presence of natural teeth on both sides of the study implant position and opposing dentition (single tooth gap).
* Patients with healed extraction sockets, which means that at implant surgery:

  * Soft tissue coverage of the socket is complete; and
  * Alveolar bone is reconsolidated (around 16 weeks after tooth extraction).

Exclusion Criteria:

* Patients with inadequate bone volume where major bone augmentation would be required at implant location.
* Inadequate anatomic situation that would prevent prosthetic-driven planning based on CBCT.
* Presence of implants neighbouring the study implant.
* Patients with inadequate oral hygiene (FMPS ≥ 20%).
* Patients with local root remnants.
* Patients with inadequate wound healing capacity.
* Patients with incomplete maxillary and mandibular growth.
* Patients with medical contraindications to implant surgery (uncontrolled bleeding disorders, psychoses, prolonged therapy-resistant functional disorders, xerostomia, weakened immune system, illnesses requiring periodic use of steroids or uncontrollable endocrine disorders.
* Patients with drug or alcohol abuse.
* Patients with allergies or hypersensitivity to zirconium oxide (ZrO2), yttrium oxide (Y2O3), hafnium dioxide (HfO2), aluminium oxide (Al2O3), and titanium (Grade 4).
* Patients with medical contraindications to implant surgery (uncontrolled bleeding disorders, psychoses, prolonged therapy-resistant functional disorders, xerostomia, weakened immune system, illnesses requiring periodic use of steroids or uncontrollable endocrine disorders).
* Patients with conditions or circumstances, in the opinion of the Investigator, which would prevent completion of study participation or interfere with analysis of study results, such as history of non-compliance or unreliability.
* Pregnancy or intention to become pregnant at any point during the study duration.

Furthermore, patients with uncontrolled periodontitis and less than 3 mm of keratinized mucosa at the day of surgery will be excluded from the study. Controlled periodontitis is defined as treated periodontitis with two or less pockets that are < 4 mm in depth or the existence of ≤ 20% bleeding on probing.

If the planned implant position is the second premolar, the adjacent molar must be present. Shortened arches with missing molars are not eligible in such a case.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2019-09-07 (Actual); Primary Completion 2025-08-29 (Estimated); Study Completion 2025-08-29 (Estimated)

PRIMARY OUTCOMES:
Bone Level Change | 12 months after implant loading (final crown restoration)
  Change in crestal bone level measured by analysis of standardized peri-apical xrays 12 months after loading [mm].

SECONDARY OUTCOMES:
Implant survival | 12 months after loading.
  Implant survival rates 3, 6 months and 1 year after loading: yes/no
14 item Oral Health Impact Profile (OHIP-14) | 12 months after loading.
  The local language version of the OPHIP-14 is a self-reported questionnaire that measures dysfunction, discomfort and disability attributed to oral conditions. The questionnaire focuses on seven dimensions of impact: Functional limitation; Pain; Psychological discomfort; Physical disability; Psychological disability; Social disability; Handicap. The patients will be asked to respond according to frequency of impact on a 5-point Likert scale coded never (score 0), hardly ever (score 1), occasionally (score 2), fairly often (score 3) and very often (score 4).

OTHER OUTCOMES:
Adverse Events | 18 months after inclusion.
  Adverse Events will be recorded at every visit.
Device Deficiencies | 18 months after inclusion.
  Any device complications and deficiencies will be recorded as Device Deficiencies.

CONTACTS AND LOCATIONS:
Locations (3):
- Dusseldorf University Hospital, Poliklinik für Zahnärztliche Prothetik, Düsseldorf, Germany
- The University of Hong Kong, Prince Philip Dental Hospital, Hong Kong, Hong Kong
- Implantology Institute, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No